CLINICAL TRIAL: NCT05618691
Title: A Double-blinded, Randomized, Placebo-controlled Study of GFH312 in Patients With Peripheral Artery Disease (PAD) and Intermittent Claudication (IC)
Brief Title: A Study of GFH312 in Patients With Peripheral Artery Disease (PAD) and Intermittent Claudication (IC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated by sponsor for reasons of adjusted clinical development strategy.
Sponsor: Zhejiang Genfleet Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Genfleet Therapeutics (Shanghai) Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GFH312X2201
Record Dates: First submitted 2022-09-15; First posted 2022-11-16 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Intermittent Claudication; Peripheral Artery Disease
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a multicenter, double-blinded, randomized, placebo-controlled study, to evaluate the safety/tolerability and efficacy in three paralleled dose groups of GFH312 compared with placebo in patients with PAD and IC.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GFH312 40mg (Experimental): Participant will receive GFH312 40mg once daily approximately at same time each day for 12 weeks.
  Interventions: Drug: GFH312
- GFH312 80mg (Experimental): Participant will receive GFH312 80mg once daily approximately at same time each day for 12 weeks.
  Interventions: Drug: GFH312
- GFH312 120mg (Experimental): Participant will receive GFH312 120mg once daily approximately at same time each day for 12 weeks.
  Interventions: Drug: GFH312
- Placebo (Experimental): Participant will receive placebo once daily approximately at same time each day for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GFH312 — Oral tablet, GFH312 will be administered at 3 dose levels, each patient in one of three groups will be given a dose of 40mg, 80mg, 120mg of the study drug.
  Arms: GFH312 120mg; GFH312 40mg; GFH312 80mg
Other: Placebo — Placebo will be administered to subjects in the placebo group
  Arms: Placebo

SUMMARY:
GFH312 could be a novel therapeutic option in the acute/chronic inflammatory process of atherosclerosis and provides potential beneficial effects to microvasculature function for PAD patients with IC in addition to preventing ischemia-reperfusion injury. This phase II study is designed to explore the clinical safety and efficacy of GFH312 after multiple oral doses, to support further development in patients with PAD or other atherosclerotic diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-80 years.
2. Patients diagnosed with PAD and IC for at least 6 months before screening and disease assessed as stage II per the Fontaine classification.
3. Patients on stable medical therapy for PAD and IC symptoms, which may include lifestyle modification (e.g., smoking cessation), a community- or home-based exercise rehabilitation program, anti-platelet medications, and individual risk factor intervention (e.g., lipid-lowering therapy, antihypertensive therapy, glycemic control) unless individually contraindicated, for at least 3 months prior to the screening visit.
4. For patients with reproductive potential, a willingness to use methods of contraception that will prevent the patients or their partners from becoming pregnant during the study.

Exclusion Criteria:

1. Participation in any clinical investigation within 4 weeks prior to enrollment or use of other investigational drugs at the time of enrollment, or within 5 half-lives at the time of enrollment, or until the expected PD effect has returned to baseline, whichever longer.
2. Patients who meet any of the following PAD related criteria:

   1. Patients with high variability in the walking distance, defined as the change ≥25% in MWD between two 6-MWT with a time interval of two to three weeks.
   2. Patients unable to hold all narcotic pain relievers for 24 hours prior to the performance of the walking test.
   3. Patients with any condition other than PAD that limits walking ability (e.g., orthopaedic disease, respiratory disease, neurological disorders).
   4. Known inflammatory disease of the arteries (other than atherosclerosis, e.g., thromboangiitis obliterans).
   5. Clinical evidence of critical limb ischemia including new or non-healing ulcers (felt secondary to critical limb ischemia), new or recent onset of resting pain in the lower extremities particularly at night (felt secondary to critical limb ischemia) and/or gangrene of the lower extremities (Fontaine stage III-IV).
   6. Patients actively attending and participating in a supervised exercise rehabilitation program (patients who have already completed such a program and remain symptomatic may be included).
3. Any of the following concomitant cardiovascular or metabolic conditions or diseases:

   1. Myocardial infarction or angina pectoris within 6 months of screening.
   2. Stroke within 3 months of screening.
   3. History of clinically significant ventricular arrhythmias, according to the discretion of the investigator, within 6 months of screening.
   4. Patients with electronic cardiac pacemaker.
   5. Significant ECG abnormalities (e.g., WPW syndrome), according to the discretion of the investigator, at screening.
   6. History of sustained and clinically significant supraventricular arrhythmias (e.g., paroxysmal atrial fibrillation/flutter) within 6 months of screening.
   7. Chronic heart failure New York Heart Association Class III or IV.
   8. Known presence of aortic aneurysm > 5 cm.
   9. Uncontrolled diabetes as defined by a random fasting glucose level of 13 mmol/L or 240 mg/dL or a HbA1c greater than 9% as measured at screening.
   10. Uncontrolled or resistant hypertension, defined as BP>160/100 mm Hg after standard anti-hypertension treatment.
4. History of unstable or severe hepatic or renal disease or another medically significant illness
5. History of any of the following chronic conditions:

   1. Malignancy of any organ system (other than localized basal or squamous cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
   2. History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result, and severe uncontrolled ulcerative colitis or Crohn's disease.
   3. History of any hypercoagulable or bleeding disorders.
   4. History of significant and active drug or alcohol abuse that could interfere with conduct of the trial within the 12 months prior to dosing. Note: investigator may establish veracity of patient history with drug or alcohol testing as deemed necessary.
6. Dementia or other mental disorders (e.g., continues to receive medication or psychological intervention) that prevent patients from following a research protocol.
7. Major surgical procedure before screening or planned to occur during the planned time frame of the study.
8. History of multiple and clinically significant recurring drug allergies.
9. Use of strong inhibitors or strong inducers of CYP3A4 within 14 days or 5 half-lives (whichever longer); or grapefruit juice or grapefruit containing products within 7 days prior to first study treatment.
10. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive HCG laboratory test.
11. Any medical condition (e.g., with a plan to receive vaccination within study duration) that in the opinion of the investigator may place the patient at higher risk from his/her participation in the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Absolute change from baseline in maximum walking distance (MWD) at Week 12 assessed by a 6-minute walking test (6-MWT) | 12 weeks
  The 6-MWT will be performed according to the 2002 American Thoracic Society Guidelines
Incidence and severity of adverse events (AEs), SAEs | 12 weeks
  Incidence and severity of adverse events (AEs), SAEs

SECONDARY OUTCOMES:
Pain-free walking distance (PFWD) at Week 12 assessed by a walking test | 12 weeks
  Pain-free walking distance would be collected during the test of 6-MWT, the 6-MWT will be performed according to the 2002 American Thoracic Society Guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- Midwest Cardiovascular Research Foundation, Davenport, Iowa, United States

IPD SHARING:
Plan to Share IPD: No